CLINICAL TRIAL: NCT01059448
Title: A Long-Term Assessment of the Safety and Efficacy of AMG 827 Subcutaneous Treatment in Subjects With Rheumatoid Arthritis
Brief Title: Safety and Efficacy of AMG 827 in Subjects With RA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy for Brodalumab in Rheumatoid Arthritis (RA)
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090402
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Amgen; RA; AMG 827; 20090061
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — brodalumab

ARMS (4):
- Placebo Q2WK / 210 mg AMG 827 Q2WK (Experimental): Participants who were administered matching placebo in parent study 20090061 and were administered 210 mg subcutaneous (SC) AMG 827 at Day 1, Week 1, Week 2, and every other week thereafter (Q2WK). Participants also continued to receive weekly intramuscular, oral or SC doses of methotrexate and folic acid or folate.
  Interventions: Drug: AMG 827
- 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (Experimental): Participants who were administered 70 mg AMG 827 in parent study 20090061 and were administered 210 mg SC AMG 827 at Day 1, Week 1, Week 2 and Q2WK thereafter. Participants also continued to receive weekly intramuscular, oral or SC doses of methotrexate and folic acid or folate.
  Interventions: Drug: AMG 827
- 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK (Experimental): Participants who were administered 140 mg AMG 827 in parent study 20090061 and were administered 210 mg SC AMG 827 at Day 1, Week 1, Week 2, and Q2WK thereafter. Participants also continued to receive weekly intramuscular, oral or SC doses of methotrexate and folic acid or folate.
  Interventions: Drug: AMG 827
- 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (Experimental): Participants who were administered 210 mg AMG 827 in parent study 20090061 and were administered 210 mg SC AMG 827 at Day 1, Week 1, Week 2, and Q2WK thereafter. Participants also continued to receive weekly intramuscular, oral or SC doses of methotrexate and folic acid or folate.
  Interventions: Drug: AMG 827

INTERVENTIONS:
Drug: AMG 827 — AMG 827 210 mg

SUMMARY:
This is an extension study for subjects who participated in Protocol 20090061 (NCT00950989). All subjects in this study will receive a 210mg injection of AMG827 for treatment for their Rheumatoid Arthritis for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent.
* Subject was randomized into study 20090061 and completed the week 16 evaluation.
* Negative test for hepatitis B virus (HBV) surface antigen, hepatitis C virus (HCV) antibody, and/or human immunodeficiency virus (HIV) in subjects if clinically indicated (eg, known recent exposure) in the opinion of the investigator.
* Subject must test negative for Tuberculosis.

Exclusion Criteria:

* Subject had any SAE reported during 20090061 that was considered to be related to IP.
* Subject is currently experiencing an infection of CTCAE grade 2 (if requiring oral antibiotics) or higher. Subject is ineligible until the infection is resolved in the opinion of the investigator.
* For subjects with > 4 weeks between the week 16 visit of 20090061 and the planned first IP dose in 20090402, subject has laboratory abnormalities at screening, including:
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT); >1.5x upper limit of normal)
* Serum total bilirubin ≥1.5 mg/dL
* Hemoglobin < 11 g/dL
* Platelet count < 125,000 /mm3
* White blood cell count < 3,000 cells/mm3
* Absolute neutrophil count < 2000/mm3
* Estimated creatinine clearance < 50 mL/min (Cockroft-Gault formula, central lab will calculate value and provide to sites)
* Subject has a significant concurrent medical conditions, including:
* Type 1 diabetes
* Poorly controlled type 2 diabetes (Hemoglobin A1c > 8.5)
* Symptomatic heart failure (New York Heart Association class II, III, or IV)
* Myocardial infarction within the last year
* Current or history of unstable angina pectoris within the last year
* Uncontrolled hypertension as defined by resting blood pressure > 150/90 mmHg prior to first IP dose (confirmed by a repeat assessment)
* Severe chronic pulmonary disease (eg, requiring oxygen therapy)
* Major chronic inflammatory disease or connective tissue disease other than rheumatoid arthritis (eg, systemic lupus erythematosus), with the exception of secondary Sjögren's syndrome
* Multiple sclerosis or any other demyelinating disease
* Active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma, or history of cancer (except successfully treated in situ cervical cancer or squamous or basal cell carcinoma of the skin)
* Any condition that, in the opinion of the investigator, might cause this study to be detrimental to the subject
* Subject is pregnant or breast feeding, or planning to become pregnant while enrolled in the study, up to the subject's last study visit including the follow-up period.
* Female subject is not willing to abstain from sexual intercourse or use 2 highly effective forms of birth control for the duration of the study and at least 40 days after the last dose (except women at least 3 years postmenopausal or surgically sterile). Highly effective methods of birth control for women include but are not limited to birth control pills, Depo Provera® injections, contraceptive implants, or occlusive cap (barrier method) in combination with barrier methods used by the man.
* Male subject is not willing to abstain from sexual intercourse or use 2 highly effective forms of birth control for the duration of the study, plus an additional 16 weeks after the last dose (except for men who are surgically sterile or whose female partners are at least 3 years postmenopausal or surgically sterile). Highly effective methods of birth control include but are not limited to a condom in combination with hormonal birth control or barrier methods used by the woman.
* Male subject (including vasectomised males) with a pregnant female partner is not willing to use effective methods to ensure that an unborn child is not exposed to AMG 827 via semen. Effective methods to ensure that an unborn child is not exposed to AMG 827 via semen include condoms or abstinence.
* Subject has used any of the following within 14 days prior to IP initiation
* Non-biologic disease-modifying anti-rheumatic drugs (DMARD) other than as allowed in 20090061
* Intra-articular, intramuscular, or intravenous corticosteroids, including adrenocorticotropic hormone
* Subject has used any of the following within 3 months prior to IP initiation
* Leflunomide
* Live vaccines
* Commercially available or experimental biologic DMARD except for AMG 827
* Subject has received gold therapy within 6 months prior to IP initiation.
* Subject received another investigational agent (other than AMG 827) or participated in an investigational device study subsequent to 20090061.
* Other investigational procedures are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2010-06-03 (Actual); Primary Completion 2011-04-05 (Actual); Study Completion 2011-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- United States (14):
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, La Jolla, California
  - Research Site, Victorville, California
  - Research Site, Sarasota, Florida
  - Research Site, Rock Island, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Grand Rapids, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Freehold, New Jersey
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Tacoma, Washington
- Bulgaria (2):
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Canada (4):
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Prague, Czechia
- Latvia (4):
  - Research Site, Bauska
  - Research Site, Daugavpils
  - Research Site, Liepāja
  - Research Site, Riga
- Mexico (5):
  - Research Site, Tijuana, Baja Calif
  - Research Site, Mexico City, Distrito F
  - Research Site, Guadalajara, Jalisco
  - Research Site, Morelia, MichoacÃ¡n
  - Research Site, San Luis Potosí City, San Luis P
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, ToruÅ"
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żyrardów
- Research Site, Merseyside, United Kingdom

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension of study 20090061 (NCT00950989). Participants were required to complete the Week 16 visit of study 2009061, sign the informed consent form, complete all screening assessments, if applicable, and meet the safety-based eligibility criteria for study 20090402.
  211 participants were enrolled across 45 centers in the United States, Canada, Czech Republic, Bulgaria, Latvia, Mexico, Poland, and the United Kingdom from 03 June 2010 to 18 May 2011.
Pre-assignment Details: 211 participants were enrolled and all 211 participants received study drug.
Period: Overall Study
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Started | 49 | 55 | 53 | 54
Completed | 0 | 0 | 0 | 0
Not Completed | 49 | 55 | 53 | 54
Not completed — Adverse Event | 1 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 4
Not completed — Disease Progression | 2 | 1 | 4 | 2
Not completed — Administrative Decision | 43 | 49 | 45 | 46
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) - All analyzable participants who were treated with at least one dose of AMG 827.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | Total
Number analyzed (Participants) | 49 | 55 | 53 | 54 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] — Measure reports age at 20090402 study baseline.
  Years | 49.9 (11.2) | 52.6 (10.7) | 54.6 (10.7) | 51.6 (8.9) | 52.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 40 | 44 | 167
  Male | 9 | 12 | 13 | 10 | 44
Race [Count of Participants; unit: Participants]
  White or Caucasian | 34 | 45 | 40 | 47 | 166
  Black or African American | 1 | 1 | 1 | 0 | 3
  Hispanic or Latino | 14 | 8 | 12 | 6 | 40
  Asian | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an event that occurred after the first dose date and before the end of study date in study 20090402; or an event that was already present prior to the initiation of the investigational product (i.e. present at study 20090402) baseline but worsened in either frequency or severity after the first dose date and before the end of study date in study 20090402.
  TEAEs also included serious treatment-emergent adverse events and clinically significant changes from baseline in hematology, chemistry and urinalysis profiles and clinically significant changes in vital sign measurements.
Time Frame: Day 1 to Week 52 of study 20090402
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 55 | 53 | 54
Participants | 28 | 32 | 31 | 32

2. Primary Outcome: Number of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response
Description: An ACR 20 response was defined as at least a 20% improvement from baseline in both tender/painful and swollen joint counts, and a 20% improvement or more in at least 3 of the following 5 criteria: physician global assessment of disease activity (PGA), subject global assessment of disease activity (SGA), participant global assessment of joint pain, participant self-assessment of disability (Health Assessment Questionnaire, HAQ-DI), and acute phase reactant: erythrocyte sedimentation rate (ESR) or C-Reactive Protein (CRP), whichever had a bigger improvement. Participants were excluded from analysis if an ACR 20 response could not be determined due to missing component data.
  Baseline refers to the baseline in parent study 20090061.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 47 | 54 | 53 | 52
Participants
  20090402 Week 2: number analyzed (Participants) | 46 | 53 | 52 | 52
  20090402 Week 2 | 21 | 24 | 26 | 24
  20090402 Week 4 | 27 | 26 | 24 | 32
  20090402 Week 8: number analyzed (Participants) | 46 | 53 | 47 | 49
  20090402 Week 8 | 27 | 31 | 27 | 29
  20090402 Week 12: number analyzed (Participants) | 38 | 46 | 43 | 40
  20090402 Week 12 | 25 | 24 | 23 | 22
  20090402 Week 16: number analyzed (Participants) | 32 | 44 | 40 | 42
  20090402 Week 16 | 19 | 28 | 23 | 22
  20090402 Week 20: number analyzed (Participants) | 29 | 33 | 29 | 33
  20090402 Week 20 | 19 | 24 | 15 | 15
  20090402 Week 24: number analyzed (Participants) | 23 | 27 | 31 | 21
  20090402 Week 24 | 12 | 17 | 17 | 12
  20090402 Week 36: number analyzed (Participants) | 12 | 13 | 13 | 14
  20090402 Week 36 | 7 | 6 | 5 | 7
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 0 |  |  |

3. Primary Outcome: Number of Participants Who Achieved an ACR 50 Response
Description: An ACR 50 response was defined as at least a 50% improvement from baseline in both tender/painful and swollen joint counts, and a 50% improvement or more in at least 3 of the following 5 criteria: PGA, SGA, participant global assessment of joint pain, participant self-assessment of disability (HAQ-DI), and acute phase reactant: ESR or CRP, whichever had a bigger improvement. Participants were excluded from analysis if an ACR 50 response could not be determined due to missing component data.
  Baseline refers to the baseline in parent study 20090061.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 47 | 54 | 53 | 52
Participants
  20090402 Week 2: number analyzed (Participants) | 47 | 53 | 52 | 52
  20090402 Week 2 | 8 | 8 | 12 | 7
  20090402 Week 4 | 8 | 10 | 10 | 10
  20090402 Week 8: number analyzed (Participants) | 46 | 54 | 47 | 49
  20090402 Week 8 | 10 | 9 | 13 | 11
  20090402 Week 12: number analyzed (Participants) | 38 | 46 | 43 | 40
  20090402 Week 12 | 13 | 10 | 10 | 10
  20090402 Week 16: number analyzed (Participants) | 33 | 44 | 40 | 42
  20090402 Week 16 | 9 | 7 | 12 | 11
  20090402 Week 20: number analyzed (Participants) | 29 | 33 | 29 | 33
  20090402 Week 20 | 9 | 10 | 5 | 8
  20090402 Week 24: number analyzed (Participants) | 22 | 27 | 31 | 21
  20090402 Week 24 | 6 | 6 | 6 | 9
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 4 | 2 | 2 | 2
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 0 |  |  |

4. Primary Outcome: Number of Participants Who Achieved an ACR 70 Response
Description: An ACR 70 response was defined as at least a 70% improvement from baseline in both tender/painful and swollen joint counts, and a 70% improvement or more in at least 3 of the following 5 criteria: PGA, SGA, participant global assessment of joint pain, participant self-assessment of disability (HAQ-DI), and acute phase reactant: ESR or CRP, whichever had a bigger improvement. Participants were excluded from analysis if an ACR 70 response could not be determined due to missing component data.
  Baseline refers to the baseline in parent study 20090061.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 54 | 53 | 52
Participants
  20090402 Week 2: number analyzed (Participants) | 47 | 53 | 52 | 52
  20090402 Week 2 | 0 | 4 | 3 | 2
  20090402 Week 4 | 2 | 4 | 3 | 2
  20090402 Week 8: number analyzed (Participants) | 47 | 54 | 47 | 49
  20090402 Week 8 | 5 | 4 | 1 | 4
  20090402 Week 12: number analyzed (Participants) | 38 | 46 | 43 | 40
  20090402 Week 12 | 5 | 5 | 2 | 2
  20090402 Week 16: number analyzed (Participants) | 33 | 44 | 40 | 42
  20090402 Week 16 | 3 | 3 | 5 | 5
  20090402 Week 20: number analyzed (Participants) | 29 | 33 | 29 | 33
  20090402 Week 20 | 4 | 3 | 1 | 1
  20090402 Week 24: number analyzed (Participants) | 23 | 27 | 31 | 21
  20090402 Week 24 | 0 | 2 | 2 | 6
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 0 | 0 | 1 | 2
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 0 |  |  |

5. Primary Outcome: Change From Baseline in Disease Activity Score 28 Joint (DAS28) Score
Description: The DAS28 is a composite score that is based on a 28-joint count (using 28 tender and 28 swollen joints), ESR, and SGA. The following formula was used where T/P28 and SW28 represent the tender and swollen 28 joint counts, respectively. The 28 joint counts include 10 proximal interphalangeal, 10 metacarpophalangeal, 2 wrist, 2 elbow, 2 shoulder, and 2 knee joints.
  DAS28 = 0.56 √T/P28 + 0.28 √SW28 + 0.7 x ln (ESR) +0.014 x SGA.
  DAS28 score ranged from 0 to 10, where a higher score represented higher disease activity. A negative change from baseline indicated a reduction in disease activity.
  Baseline refers to the baseline in parent study 20090061.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least 1 dose of AMG 827.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 46 | 54 | 53 | 52
Score on a Scale
  20090402 Week 2: number analyzed (Participants) | 45 | 53 | 52 | 52
  20090402 Week 2 | -1.60 (1.02) | -1.39 (1.26) | -1.49 (1.22) | -1.31 (1.07)
  20090402 Week 4: number analyzed (Participants) | 45 | 54 | 53 | 52
  20090402 Week 4 | -1.60 (1.30) | -1.54 (1.32) | -1.40 (1.18) | -1.46 (1.08)
  20090402 Week 8: number analyzed (Participants) | 46 | 53 | 47 | 49
  20090402 Week 8 | -1.69 (1.32) | -1.65 (1.40) | -1.50 (1.12) | -1.64 (1.25)
  20090402 Week 12: number analyzed (Participants) | 37 | 46 | 43 | 40
  20090402 Week 12 | -1.99 (1.08) | -1.81 (1.29) | -1.38 (1.39) | -1.46 (1.15)
  20090402 Week 16: number analyzed (Participants) | 32 | 44 | 40 | 42
  20090402 Week 16 | -2.05 (1.27) | -1.71 (1.20) | -1.63 (1.37) | -1.53 (1.27)
  20090402 Week 20: number analyzed (Participants) | 27 | 32 | 29 | 33
  20090402 Week 20 | -1.94 (1.35) | -1.70 (1.26) | -1.61 (1.04) | -1.52 (1.21)
  20090402 Week 24: number analyzed (Participants) | 22 | 27 | 31 | 21
  20090402 Week 24 | -1.85 (1.00) | -1.66 (1.12) | -1.49 (1.21) | -1.99 (1.38)
  20090402 Week 36: number analyzed (Participants) | 12 | 13 | 13 | 14
  20090402 Week 36 | -1.87 (1.30) | -1.60 (1.01) | -1.61 (1.35) | -1.77 (1.46)
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 0.18 (NA) — Only 1 participant had evaluable data, therefore, standard deviation could not be calculated |  |  |

6. Primary Outcome: Number of Participants With a DAS28 Score < 2.6
Description: The DAS28 is a composite score that is based on a 28-joint count (using 28 tender and 28 swollen joints), ESR, and SGA. The following formula was used where T/P28 and SW28 represent the tender and swollen 28 joint counts, respectively. The 28 joint counts include 10 proximal interphalangeal, 10 metacarpophalangeal, 2 wrist, 2 elbow, 2 shoulder, and 2 knee joints.
  DAS28 = 0.56 √T/P28 + 0.28 √SW28 + 0.7 x ln (ESR) +0.014 x SGA.
  DAS28 score ranged from 0 to 10, where a higher score represented higher disease activity. A score of <2.6 indicated disease activity remission.
  1 participant in the Arm "Placebo Q2WK / 210 mg AMG 827 Q2WK" was missing baseline data for DAS28.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 55 | 53 | 54
Participants
  Parent Study 20090061 Baseline: number analyzed (Participants) | 48 | 55 | 53 | 54
  Parent Study 20090061 Baseline | 0 | 0 | 0 | 0
  20090402 Baseline | 2 | 2 | 0 | 2
  20090402 Week 2: number analyzed (Participants) | 46 | 53 | 52 | 52
  20090402 Week 2 | 0 | 3 | 1 | 1
  20090402 Week 4: number analyzed (Participants) | 46 | 54 | 53 | 52
  20090402 Week 4 | 1 | 4 | 1 | 1
  20090402 Week 8: number analyzed (Participants) | 47 | 53 | 47 | 49
  20090402 Week 8 | 1 | 3 | 0 | 5
  20090402 Week 12: number analyzed (Participants) | 38 | 46 | 43 | 40
  20090402 Week 12 | 2 | 6 | 0 | 1
  20090402 Week 16: number analyzed (Participants) | 33 | 44 | 40 | 42
  20090402 Week 16 | 1 | 4 | 1 | 5
  20090402 Week 20: number analyzed (Participants) | 28 | 32 | 29 | 33
  20090402 Week 20 | 1 | 2 | 1 | 1
  20090402 Week 24: number analyzed (Participants) | 23 | 27 | 31 | 21
  20090402 Week 24 | 0 | 1 | 1 | 2
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 0 | 1 | 1 | 1
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 0 |  |  |

7. Primary Outcome: DAS28 Score at All Measured Timepoints
Description: The DAS28 is a composite score that is based on a 28-joint count (using 28 tender and 28 swollen joints), ESR, and SGA. The following formula was used where T/P28 and SW28 represent the tender and swollen 28 joint counts, respectively. The 28 joint counts include 10 proximal interphalangeal, 10 metacarpophalangeal, 2 wrist, 2 elbow, 2 shoulder, and 2 knee joints.
  DAS28 = 0.56 √T/P28 + 0.28 √SW28 + 0.7 x ln (ESR) +0.014 x SGA.
  DAS28 score ranged from 0 to 10, where a higher score represented higher disease activity.
  1 participant in the Arm "Placebo Q2WK / 210 mg AMG 827 Q2WK" was missing baseline data for DAS28.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 55 | 53 | 54
Score on a Scale
  Parent Study 20090061 Baseline: number analyzed (Participants) | 48 | 55 | 53 | 54
  Parent Study 20090061 Baseline | 6.52 (0.85) | 6.40 (0.78) | 6.45 (0.81) | 6.41 (0.72)
  20090402 Baseline | 5.16 (1.43) | 5.22 (1.30) | 5.33 (1.17) | 5.49 (1.38)
  20090402 Week 2: number analyzed (Participants) | 46 | 53 | 52 | 52
  20090402 Week 2 | 4.97 (1.22) | 5.00 (1.32) | 4.96 (1.30) | 5.09 (1.27)
  20090402 Week 4: number analyzed (Participants) | 46 | 54 | 53 | 52
  20090402 Week 4 | 5.00 (1.41) | 4.87 (1.29) | 5.06 (1.23) | 4.96 (1.30)
  20090402 Week 8: number analyzed (Participants) | 47 | 53 | 47 | 49
  20090402 Week 8 | 4.81 (1.34) | 4.75 (1.33) | 4.97 (1.23) | 4.79 (1.48)
  20090402 Week 12: number analyzed (Participants) | 38 | 46 | 43 | 40
  20090402 Week 12 | 4.64 (1.17) | 4.59 (1.34) | 5.13 (1.32) | 5.02 (1.25)
  20090402 Week 16: number analyzed (Participants) | 33 | 44 | 40 | 42
  20090402 Week 16 | 4.61 (1.23) | 4.62 (1.17) | 4.93 (1.38) | 4.94 (1.49)
  20090402 Week 20: number analyzed (Participants) | 28 | 32 | 29 | 33
  20090402 Week 20 | 4.58 (1.29) | 4.52 (1.27) | 4.73 (1.12) | 4.98 (1.33)
  20090402 Week 24: number analyzed (Participants) | 23 | 27 | 31 | 21
  20090402 Week 24 | 4.71 (1.08) | 4.61 (1.13) | 4.94 (1.19) | 4.57 (1.61)
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 4.66 (1.13) | 4.54 (1.15) | 5.06 (1.26) | 4.90 (1.56)
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 7.93 (NA) — Only 1 participant had evaluable data, therefore, standard deviation could not be calculated |  |  |

8. Primary Outcome: CRP Levels at All Measured Timepoints
Description: All blood samples were taken before the dose of IP was administered. Blood samples were processed and sent to the central laboratory. The central laboratory were responsible for completing assessments.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 55 | 53 | 54
Milligrams per Liter (mg/L)
  Parent Study 20090061 Baseline | 12.95 (11.99) | 14.74 (17.50) | 18.91 (24.35) | 12.22 (10.69)
  20090402 Baseline: number analyzed (Participants) | 49 | 55 | 52 | 54
  20090402 Baseline | 11.42 (12.13) | 12.23 (12.75) | 14.48 (18.84) | 12.25 (12.49)
  20090402 Week 2: number analyzed (Participants) | 45 | 52 | 52 | 52
  20090402 Week 2 | 9.67 (8.91) | 10.44 (10.31) | 18.58 (28.49) | 10.56 (11.04)
  20090402 Week 4: number analyzed (Participants) | 49 | 54 | 52 | 51
  20090402 Week 4 | 10.70 (10.05) | 12.79 (15.91) | 14.46 (15.39) | 11.47 (11.67)
  20090402 Week 8: number analyzed (Participants) | 47 | 53 | 46 | 49
  20090402 Week 8 | 9.18 (10.51) | 12.19 (14.18) | 13.84 (15.62) | 13.20 (15.11)
  20090402 Week 12: number analyzed (Participants) | 39 | 47 | 43 | 40
  20090402 Week 12 | 9.07 (9.38) | 12.61 (14.61) | 15.68 (14.82) | 14.54 (13.25)
  20090402 Week 16: number analyzed (Participants) | 33 | 43 | 40 | 42
  20090402 Week 16 | 12.09 (12.69) | 12.91 (20.22) | 16.01 (17.40) | 12.92 (11.70)
  20090402 Week 20: number analyzed (Participants) | 29 | 32 | 29 | 33
  20090402 Week 20 | 10.21 (12.13) | 10.59 (12.05) | 14.14 (16.69) | 14.79 (18.38)
  20090402 Week 24: number analyzed (Participants) | 22 | 28 | 31 | 21
  20090402 Week 24 | 7.99 (5.82) | 8.76 (9.16) | 16.50 (21.01) | 9.41 (10.04)
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 8.49 (9.96) | 9.92 (12.22) | 12.02 (17.38) | 8.89 (8.71)
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 22.10 (NA) — Only 1 participant had evaluable data, therefore, standard deviation could not be calculated |  |  |

9. Primary Outcome: ESR at All Measured Timepoints
Description: All blood samples were taken before the dose of IP was administered. ESR was performed locally at each site and the ESR data was submitted to the central laboratory.
Time Frame: Baseline of parent study 20090061 to Week 2, 4, 8, 12, 16, 20, 24, 36 and 48 of study 20090402.
Population: FAS - All analyzable participants who were treated with at least one dose of AMG 827.
Measure: Mean (Standard Deviation); unit: millimeters per hour (mm/hr)
Arm/Group | Placebo Q2WK / 210 mg AMG 827 Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Number analyzed (Participants) | 49 | 55 | 53 | 54
millimeters per hour (mm/hr)
  Parent Study 20090061 Baseline | 50.12 (20.53) | 44.27 (18.72) | 45.81 (21.97) | 45.06 (20.03)
  20090402 Baseline | 38.35 (27.78) | 38.15 (23.79) | 41.89 (22.27) | 39.15 (24.70)
  20090402 Week 2: number analyzed (Participants) | 46 | 53 | 52 | 52
  20090402 Week 2 | 36.78 (21.43) | 36.83 (27.11) | 37.65 (19.24) | 37.00 (25.23)
  20090402 Week 4: number analyzed (Participants) | 49 | 54 | 53 | 52
  20090402 Week 4 | 39.27 (23.73) | 36.07 (21.44) | 40.53 (23.50) | 38.31 (24.70)
  20090402 Week 8: number analyzed (Participants) | 47 | 54 | 47 | 49
  20090402 Week 8 | 37.40 (23.26) | 34.65 (23.14) | 38.43 (19.50) | 35.55 (23.52)
  20090402 Week 12: number analyzed (Participants) | 39 | 47 | 43 | 40
  20090402 Week 12 | 36.31 (18.30) | 36.09 (24.30) | 42.28 (22.74) | 39.30 (22.54)
  20090402 Week 16: number analyzed (Participants) | 33 | 44 | 40 | 42
  20090402 Week 16 | 38.21 (23.08) | 40.27 (26.07) | 43.78 (23.23) | 39.43 (22.81)
  20090402 Week 20: number analyzed (Participants) | 29 | 32 | 29 | 33
  20090402 Week 20 | 43.41 (28.27) | 35.16 (24.73) | 38.00 (26.25) | 40.48 (26.71)
  20090402 Week 24: number analyzed (Participants) | 23 | 28 | 31 | 21
  20090402 Week 24 | 42.83 (25.05) | 41.07 (23.14) | 40.58 (21.12) | 42.62 (27.23)
  20090402 Week 36: number analyzed (Participants) | 13 | 13 | 13 | 14
  20090402 Week 36 | 36.62 (16.19) | 38.69 (23.22) | 36.85 (18.07) | 38.07 (26.39)
  20090402 Week 48: number analyzed (Participants) | 1 | 0 | 0 | 0
  20090402 Week 48 | 65.00 (NA) — Only 1 participant had evaluable data, therefore, standard deviation could not be calculated |  |  |

ADVERSE EVENTS:
Time Frame: From first dose of study drug in 20090402 until the end of study (maximum duration was 366 days)
Groups:
- Placebo / AMG 827 210 mg Q2WK: Participants who were administered matching placebo in parent study 2009061 and were administered 210 mg subcutaneous (SC) AMG 827 at Day 1, Week 1, Week 2, and every other week thereafter (Q2WK).
  Participants also received weekly intramuscular, oral or SC doses of methotrexate.
Arm/Group | Placebo / AMG 827 210 mg Q2WK | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK
Serious Adverse Events (participants affected / at risk) | 2/49 | 5/55 | 1/53 | 0/54
Other Adverse Events (participants affected / at risk) | 15/49 | 18/55 | 19/53 | 22/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo / AMG 827 210 mg Q2WK (N=49) | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (N=55) | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK (N=53) | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (N=54)
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo / AMG 827 210 mg Q2WK (N=49) | 70 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (N=55) | 140mg AMG 827 Q2WK / 210mg AMG 827 Q2WK (N=53) | 210 mg AMG 827 Q2WK / 210 mg AMG 827 Q2WK (N=54)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 3
Conjunctivitis (Eye disorders) | 0 | 3 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 3
Injection site pain (General disorders) | 5 | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 4 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 7 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 3
Headache (Nervous system disorders) | 1 | 4 | 3 | 2

LIMITATIONS AND CAVEATS:
The study was terminated on 18 May 2011 because AMG 827 was not shown to be efficacious in the parent study (Study 20090061) when compared to placebo at any dose as measured by ACR 20, 50, or 70 responses. In addition, there was no observed difference compared to placebo in responses as measured by the individual components of the ACR response criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.